CLINICAL TRIAL: NCT01246258
Title: Otolith Function in Patients With Primary Ciliary Dyskinesia: a Pilot Study
Brief Title: Otolith Function in Patients With Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: JROHH0046
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2014-08

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: primary ciliary dyskinesia; otolith; vestibular tests
MeSH Terms: conditions — Ciliary Motility Disorders | interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Test group: Standard tests of balance function
  Interventions: Other: Vestibular evoked myogenic potentials (VEMPs); Other: Utricular centrifugation test

INTERVENTIONS:
Other: Vestibular evoked myogenic potentials (VEMPs) — Standard test of balance function
Other: Utricular centrifugation test — Standard test of balance function

SUMMARY:
The purpose of this study is to determine whether patients with primary ciliary dyskinesia (PCD) have reduced or absent otolith function.The otolith system is a specific part of the inner ear vestibular (balance) system that detects linear movement.

DETAILED DESCRIPTION:
Primary ciliary dyskinesia (PCD) is a genetically inherited condition. It is due to structural abnormalities of cilia, which are microscopic hairs found in organs and cells throughout the body. Patients with this condition typically develop upper respiratory tract symptoms such as sinusitis and glue ear, lower respiratory tract problems such as recurrent chest infections, and fertility problems. There is currently no evidence that patients with PCD have a higher incidence of balance problems. However, recent animal studies have shown that cilia may also be important in the development of part of the inner ear balance (vestibular) system, specifically the part that detects linear movement known as the otolith system.

The investigators hope to determine whether patients with PCD have absent or reduced otolith function compared to the normal population. Balance problems are not currently screened for in PCD patients, and could be unrecognized and therefore untreated. It is also possible that PCD patients have compensated for absent otolith function and so are unaffected under normal circumstances; any additional insult to their balance system would cause more pronounced difficulties than expected and treatment might need to reflect this.

ELIGIBILITY:
Inclusion Criteria:

* aged 16-30 years
* Confirmed diagnosis of PCD under the care of the PCD team at the Royal Brompton Hospital

Exclusion Criteria:

* Aged under 16 years
* Unconfirmed or "suspected" PCD
* Previous history of balance disorders or diagnoses
* Previous history of sensorineural hearing loss
* Previous middle or inner ear surgery (other than grommet insertion)

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ten patients from the PCD clinic at the Royal Brompton Hospital, London.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Rimmer, MA FRCS, Principal Investigator — Imperial College Healthcare NHS Trust; Jonny Harcourt, MA FRCS, Study Director — Imperial College Healthcare NHS Trust
Locations (1):
- Charing Cross Hospital, London, United Kingdom

REFERENCES:
- [Result] Rimmer J, Patel M, Agarwal K, Hogg C, Arshad Q, Harcourt J. Peripheral vestibular dysfunction in patients with primary ciliary dyskinesia: abnormal otoconial development? Otol Neurotol. 2015 Apr;36(4):662-9. doi: 10.1097/MAO.0000000000000592. PMID 25226371

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: Utricular centrifugation and VEMPs: Standard tests of balance function
Period: Overall Study
Arm/Group | Test Group
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Vestibular Evoked Myogenic Potentials (VEMPs)
Description: These are the balance tests that specifically assess the otolith organ.
Time Frame: one day
Measure: Number; unit: participants
Groups:
- Test Group: VEMPs
Arm/Group | Test Group
Number analyzed (Participants) | 5
participants
  Normal VEMP | 0
  Reduced/absent VEMP bilaterally | 3
  Reduced/absent VEMP unilaterally | 2

2. Other Pre Specified Outcome: Utricular Centrifugation Test (UCF)
Description: balance assessment
Time Frame: one day
Measure: Number; unit: participants
Arm/Group | Test Group
Number analyzed (Participants) | 5
participants
  Normal UCF | 2
  Asymmetrical UCF (not significant) | 3
  Pathological UCF asymmetry | 0

ADVERSE EVENTS:
Arm/Group | Test Group
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes